CLINICAL TRIAL: NCT06305533
Title: Efficacy of Photodynamic Therapy and LASER Disinfection as Adjunct to Nonsurgical Periodontal Therapy for Treatment of Periodontitis: Randomized Clinical Trial
Brief Title: Efficacy of Photodynamic Therapy and LASER Disinfection in Periodontal Therapy for Treatment of Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Zahraa Talib Abid, Dentist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 854623
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: This study is 3 arm, split-mouth, double blinded, randomized clinical trial. The first group will receive RSD only, the second group will be treated with RSD + aPDT with ICG as a PS, and the last group will receive RSD + Laser disinfection.
Who Masked: Outcomes Assessor
Masking Description: Sites will randomly be assigned to test or control groups according to a computer-generated list. Allocation concealment will be assured by opaque, sealed envelopes prepared and sequentially numbered by a person not otherwise involved in the study. The person responsible for delivering treatment will be aware about allocation of the groups, while the assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Root surface debridement only
  Interventions: Procedure: Root surface debridement
- Test group 1 (Biolase group) (Active Comparator): Root surface debridement and laser disinfection, the diode Laser (Bolas) will be used to disinfect the inner layer of the pockets and thus reducing the microbial load.
  Interventions: Device: LASER disinfection; Procedure: Root surface debridement
- Test group 2 (Quicklase group) (Active Comparator): Root surface debridement and photodynamic therapy using a Indocyanine green photosensitizer activated with diode laser (Quicklase)
  Interventions: Device: Photodynamic therapy; Procedure: Root surface debridement

INTERVENTIONS:
Device: LASER disinfection — In test group 1, the diode Laser will be used to disinfect the inner layer of the pockets and thus reducing the microbial load. Diode laser (Biolase, EpicX, BIOLASE, Inc, USA) settings will be as follows: wavelength: 940nm; power: 1W; 300μm uninitiated fibers; continuous radiation mode; and energy level: 80 J/s. The laser fibers then will be inserted into the pockets in such a way that they will be in contact with the soft tissue wall of the pockets and parallel to the root surface and then will be moved to the apical surface through a horizontal sweeping motion (1mm/s) while remaining in contact with the soft tissue wall of the pockets.
  Arms: Test group 1 (Biolase group)
Device: Photodynamic therapy — the second test group will receive additional adjunctive aPDT using a ICG photosensitizer activated with diode laser. In details, pockets will be irrigated by a syringe loaded with an ICG photosensitizer solution (Verdye, Diagnostic green, Germany) at a concentration of 5mg/ml. The ICG solution will be allowed to stay in the pockets for 2min, and washing out excess solution from the pockets before laser irradiation. Afterwards, a 300μm bulb optical fibre of the 810nm diode laser unit (QuickLase, United Kingdom) set at 300mw in pulsed mode (100ms ON/100ms OFF) will be inserted along the pocket and activated for 30s with continuous vertical movements from the bottom of the pocket to the gingival margin
  Arms: Test group 2 (Quicklase group)
Procedure: Root surface debridement — For all groups, sites with initial PPD 4-6 mm will be treated with RSD using area specific (Graecy) curettes.

SUMMARY:
The goal of this clinical trial is to Investigate the clinical and microbiological efficacies of Laser disinfection and ICG-mediated aPDT as adjunct to RSD for patients with periodontitis. The main question it aims to answer is:

Does the use of laser disinfection or ICG-mediated aPDT as adjunct to RSD are effective in improving clinical parameters and reducing the load of periodontal pathogens.

Participants will undergo full-mouth supragingival debridement by using ultrasonic device at baseline.

All patients will be instructed to brush their teeth twice daily and will be supplied with the same type of tooth paste and toothbrush, with suitable interdental aids.

All the patients will be instructed to attend again after 7 days. One week later, sites randomly allocated to control (Ctrl) group and test groups which will receive, in addition to RSD, either aPDT or periodontal pocket disinfection (Biolase). For all groups, sites with initial PPD 4-6 mm will be treated with RSD using area specific (Graecy) curettes.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (>18 years), non-smoker, with no history of any systemic disease such as diabetes mellitus. Additionally, subjects are not currently under active periodontal therapy or joining other trial in the last 3 months. All patients must be diagnosed with generalized periodontitis with at least 3 teeth in three different sextants (Anterior teeth and premolars) with 4-6 mm PPD and positive BOP. Periodontitis cases will be defined by presence of interdental CAL affecting ≥2 non adjacent teeth or if CAL at buccal/lingual aspects associated with PPD >4mm at ≥2 teeth.

Exclusion Criteria:

* Patients will be excluded if they were not diagnosed with periodontitis, smokers, those consuming antibiotics, regular user of nonsteroidal anti-inflammatory drugs, or receiving periodontal treatment 3-months prior to the study. Additionally, pregnant or mothers in a breastfeeding period, and those not willing to participate will be also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Probing Pocket Depth (PPD) | over a period of 3 months.
  PPD will be measured from the gingival margin to the base of the pocket using UNC-15 periodontal probe and the measurements in millimetre .

SECONDARY OUTCOMES:
Bleeding on probing (BOP) | over a period of 3 months.
  The BOP will be scored as 0 (absent) and 1 (present) after probing within 30s by quadrant using UNC-15 periodontal probe .
Plaque index (PI) | over a period of 3 months.
  Biofilm will be determined using a dichotomous scoring system as presence (1) or absence (0). Disclosing solution will be used to assess agreement on scoring of biofilm.
Clinical attachment loss (CAL) | over a period of 3 months.
  CAL will be measured from the cementoenamel junction to the base of the pocket using UNC-15 periodontal probe and the measurements in millimetre .
Change in bacterial load of F. nucleatum and Fretibacterium fastidiosum | over a period of 3 months.
  Real time PCR will be used to assess the detection of the following periodontal pathogens in the subgingival biofilm samples: F. nucleatum and F. fastidiosum, according to manufacturer's instructions. Identification of target bacteria through PCR will be executed using species specific primers.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided